CLINICAL TRIAL: NCT02330965
Title: Mechanistic Studies of Phase III Trial With BAF312 in Secondary Progressive Multiple Sclerosis (AMS04)
Brief Title: Mechanistic Studies of Phase III Trial With BAF312 in Secondary Progressive Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Autoimmunity Centers of Excellence (Other); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: DAIT AMS04
Record Dates: First submitted 2014-12-31; First posted 2015-01-05 (Estimated); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Secondary Progressive Multiple Sclerosis
Keywords: autoimmunity; clinical research; mechanistic studies; blood draw; cerebrospinal fluid (CSF) by lumbar puncture (optional)
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Autoimmune Diseases | interventions — Blood Specimen Collection; Phlebotomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood & Cerebrospinal Fluid Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects Assigned to BAF312: Patients with secondary progressive multiple sclerosis (SPMS) randomized to receive BAF312 (siponimod). Refer to ClinicalTrials.gov record NCT01665144 for more information.
  Interventions: Procedure: Blood Draw; Procedure: CSF collection by lumbar puncture (Optional)
- Subjects Assigned to Placebo (Controls): Patients with secondary progressive multiple sclerosis (SPMS) randomized to receive placebo. Refer to ClinicalTrials.gov record NCT01665144 for more information.
  Interventions: Procedure: Blood Draw; Procedure: CSF collection by lumbar puncture (Optional)

INTERVENTIONS:
Procedure: Blood Draw — Blood draws (65 mLs [~4 tablespoons] per blood draw) at 4 time points: Prior to study medication initiation, and at +6, +12 and+24 months post treatment initiation.
  Other Names: Phlebotomy; Venipuncture
Procedure: CSF collection by lumbar puncture (Optional) — For participants who volunteer to donate CSF samples: up to 25 mLs (<2 tablespoons): prior to study medication initiation, and at month 24 post treatment initiation.
  Other Names: CSF by LP; cerebrospinal fluid collected by lumbar puncture

SUMMARY:
The primary goal of this study is to evaluate the effects of BAF312 (siponimod) on select immune and neuronal (nerve) cells by examining laboratory specimens (blood and/or spinal fluid) at multiple time points, prior to, and following the initiation of BAF312 or placebo treatment, in patients with Secondary Progressive Multiple Sclerosis (SPMS) who are enrolled in a clinical trial (NCT01665144) to evaluate the effectiveness and safety of BAF312.

DETAILED DESCRIPTION:
This study is complementary to a multi-center, randomized, double-blind,parallel-group, placebo-controlled, variable treatment duration study comparing the efficacy and safety of BAF312 to placebo in patients with SPMS (NCT01665144). Investigators will explore both immunological and neuroprotective mechanisms of BAF312 (siponimod), a novel agent in the setting of a SPMS clinical trial.

This study is part of a multi-center study, with the University of Michigan serving as the central site.

ELIGIBILITY:
Inclusion Criteria:

* Participants enrolled in the multicenter, randomized, double-blind, parallel-group, placebo-controlled, variable treatment duration study comparing the efficacy and safety of BAF312 to placebo in patients with Secondary Progressive Multiple Sclerosis (SPMS) Protocol No. CBAF312A2304 (sponsored by Novartis). Refer to ClinicalTrials.gov record NCT01665144.
* Subjects enrolled at one of the participating AMS04 study sites located in the United States.
* Subject must be able to provide written informed consent.

Exclusion Criteria:

* Subjects with severe bleeding disorders, platelet count less than (<)50,000/microliters (μL), and/or who are currently on full anticoagulant therapy will be excluded from the optional CSF collections.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Ambulatory participants with Secondary Progressive Multiple Sclerosis (SPMS) enrolled in the EXPAND trial (BAF312 treated and placebo [control] participants) may be enrolled in this study after the EXPAND baseline visit has occurred provided that the subject has not passed the Month 12 time point.
  -Refer to ClinicalTrials.gov record NCT01665144.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2014-12; Primary Completion 2017-07-12 (Actual); Study Completion 2017-07-12 (Actual)

PRIMARY OUTCOMES:
Change in frequency of MBP-reactive Th17 cells | From baseline to the follow-up time points (Open label phase + 6 months and OLP +12 months).
  Evaluation (BAF312 versus placebo) of dominant cytokines produced by myelin basic protein (MBP)-stimulated peripheral blood mononuclear cells (PBMCs), measured by ELISpot.

SECONDARY OUTCOMES:
Change in frequency of polyclonal CD4+ Th17, Th1, Th2, and Treg cells | From baseline to the follow-up time points (Open label phase + 6 months and OLP +12 months).
  Compare BAF312 and Placebo (Control) Groups
Change in chemokine and cytokines levels | From baseline to the follow-up time points (Open label phase + 6 months and OLP +12 months).
  Compare BAF312 and Placebo (Control) Groups
Change in Regulatory B Cells | From baseline to the follow-up time points (Open label phase + 6 months and OLP +12 months).
  Compare BAF312 and Placebo (Control) Groups
Changes of clinical status and lymphocyte subgroups | From baseline to the follow-up time points (Open label phase + 6 months and OLP +12 months).
  Compare BAF312 and Placebo (Control) Groups

CONTACTS AND LOCATIONS:
Overall Officials: Yang Mao-Draayer, MD, PhD, Study Chair — Multiple Sclerosis Center - University of Michigan Health System; David Fox, MD, Study Chair — Division of Rheumatology - University of Michigan Health System
Locations (13):
- United States (13):
  - Jordan Research & Education Institute: Sutter Alta Bates Summit, Berkeley, California
  - University of Southern California, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - University of Colorado, Aurora, Colorado
  - University of Michigan Health System -Multiple Sclerosis Center, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - University of New Mexico: Health Sciences Center, Albuquerque, New Mexico
  - South Shore Neurologic Associates - Multiple Sclerosis Care Center, Patchogue, New York
  - Carolinas Medical Center (CMC), Charlotte, North Carolina
  - Cleveland Clinic: Mellen Center for Multiple Sclerosis, Cleveland, Ohio
  - Providence Multiple Sclerosis Center, Portland, Oregon
  - Swedish Neuroscience Institute, Seattle, Washington

REFERENCES:
- [Result] Wu Q, Mills EA, Wang Q, Dowling CA, Fisher C, Kirch B, Lundy SK, Fox DA, Mao-Draayer Y; AMS04 Study Group. Siponimod enriches regulatory T and B lymphocytes in secondary progressive multiple sclerosis. JCI Insight. 2020 Feb 13;5(3):e134251. doi: 10.1172/jci.insight.134251. PMID 31935197
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Relevant Clinical Trials.gov Record: NCT01665144 — http://clinicaltrials.gov/ct2/show/record/NCT01665144?term=BAF312&rank=4